CLINICAL TRIAL: NCT02300571
Title: An Observational Retrospective/Prospective Study of the Combination of Post-transplant High Dose Cyclophosphamide, Tacrolimus and Mycophenolate Mofetil for the Prevention of Acute Graft-versus-Host Disease in Patients Eligible to Allogeneic Hematopoietic Stem Cell Transplant Using Peripheral Blood Stem Cells (PBSC) From Unrelated or Related, HLA-identical or Partially Mismatched Donors
Brief Title: Observational Study of the Combination of Post-transplant High Dose Cyclophosphamide, Tacrolimus and Mycophenolate Mofetil for the Prevention of Acute Graft-versus-Host Disease in Patients Eligible to Allogeneic Hematopoietic Stem Cell Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: HDCTX 2013
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study is proposed to observe the effect of high-dose, post-transplantation cyclophosphamide after a T cell-replete, HLA-matched PBSC graft from an HLA-identical or mismatched donor.

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation (HCT) remains the only curative approach for many hematological malignancies. In allogeneic HCT the donor immune system through the donor lymphocytes exerts both a beneficial and detrimental effect. Graft versus host disease (GVHD) represents the major complication and cause of mortality of allogeneic HCT. The principal aim that clinical transplant research must accomplish in the next years is to elaborate a transplant strategy devoid of any GVHD but still capable of generating, through donor lymphocytes, the graft versus tumor effect (GVT). The most used GVHD prophylaxis regimen remains the association of a calcineurin-inhibitor (CNIs) for six months and four low-doses of methotrexate (MTX) but the long length prophylaxis impacts on the process of post-transplant immune reconstitution slowing it down and exposing patients to a high risk of developing severe infections. The use of post-transplant cyclophosphamide looks the most promising among the new approaches to GVHD control. The study design is an observational retrospective/prospective Study in Patients Eligible to Allogeneic Hematopoietic Stem Cell Transplant using Peripheral Blood Stem Cells (PBSC) from unrelated or related, HLA-identical or partially mismatched donors. In case of unrelated donor, donor selection will be done accordingly to Italian Bone Marrow Donor Registry (IBMDR). This protocol and the treatment plan outlined below are limited to the plan or GVHD prevention.

The treatment plan for all patients including pre-conditioning therapy, TBI/chemotherapy, central nervous system prophylaxis and other planned therapies, is described in the primary transplant protocols which the patient has been assigned by the investigational site.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled for transplant of 'mobilized' peripheral blood stem cells (PBSC) from a genotypically HLA-unrelated or related identical or partially mismatched stem cell donor.
2. Patient is ≥ 18 years and ≤ 65 years of age.
3. Diagnosis of malignancy. Patients will be divided on the basis of their disease in low risk and high risk patients.

   High risk diseases: AML > CR1, ALL > CR1, CML in CP #2, AP or BP, non-Hodgkin's lymphoma > CR2, Hodgkin's lymphoma > CR2, other patient with refractory malignancy Low risk: multiple myeloma (all patients), AML in CR1, myelodysplastic syndrome beyond RA (including CMML) and ALL in CR1.
4. Patient or legal guardian has signed/dated the informed consent form.
5. Female patients must have a negative pregnancy test (blood or urine) unless they are prepuberal or surgically sterile.
6. Estimated Creatinine Clearance ≥ 60 mL/min at time of consent.
7. Total bilirubin is ≤ 1.5 times the upper limit of normal at time of consent.
8. SGOT and SGPT are ≤ 2.0 times the upper limit of normal at time of consent.

Exclusion Criteria:

1. Patient > 65 years of age
2. Patient has not signed/dated the informed consent form.
3. Patient is receiving a T-cell depleted hematopoietic stem cell graft.
4. Pregnant or lactating women
5. Patient has an acute pulmonary infection suspected on the basis of abnormal chest x-ray.
6. Patient has an active systemic infection not controlled with anti-microbial therapy.
7. Patient is a known carrier of any of the Human Immune Deficiency Viruses (HIV-1 or others).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Hematological Malignancies Eligible to Allogeneic Hematopoietic Stem Cell Transplant using Peripheral Blood Stem Cells (PBSC) from unrelated or related, HLA-identical or partially mismatched donors
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the observed GVHD rate and infections | 100 day
  Evaluations through day 100 after transplantation will be performed with:
  1. Complete blood count (CBC), including differential and platelet count per standard practice guidelines at the performance site.
  2. Blood chemistries: including sodium, potassium, chloride, bicarbonate (HCO3) or total carbon dioxide (CO2), glucose, blood urea nitrogen (BUN), creatinine, calcium, magnesium, phosphorus, total bilirubin, total protein, albumin, serum glutamic oxaloacetic transaminase (SGOT), lactic dehydrogenase (LDH), alkaline phosphatase per standard practice guidelines at the performance site.
  Tacrolimus whole blood concentrations weekly starting on day 6. CMV surveillance, Aspergillus surveillance will be performed per standard practice guidelines at the performance site.
  Evaluations after 100 days post-transplant will be completed per standard practice guidelines at each performance site.

SECONDARY OUTCOMES:
Overall survival | 1 years
  To determine the overall survival at 1 years (OS)
Progression-free survival | 1 years
  To determine progression-free survival at 1 years (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Aglietta, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia; Franca Fagioli, MD, Study Chair — Ospedale Regina Margherita; Fabrizio Carnevale-Schianca, MD, Study Chair — Fondazione del Piemonte per l'Oncologia
Locations (2):
- Italy (2):
  - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Ospedale Regina Margherita, Torino

REFERENCES:
- [Derived] Carnevale-Schianca F, Caravelli D, Gallo S, Becco P, Paruzzo L, Poletto S, Polo A, Mangioni M, Salierno M, Berger M, Pessolano R, Saglio F, Gottardi D, Rota-Scalabrini D, Grignani G, Fizzotti M, Ferrero I, Frascione PMM, D'Ambrosio L, Gaidano V, Gammaitoni L, Sangiolo D, Saglietto A, Vassallo E, Cignetti A, Aglietta M, Fagioli F. Post-Transplant Cyclophosphamide and Tacrolimus-Mycophenolate Mofetil Combination Governs GVHD and Immunosuppression Need, Reducing Late Toxicities in Allogeneic Peripheral Blood Hematopoietic Cell Transplantation from HLA-Matched Donors. J Clin Med. 2021 Mar 11;10(6):1173. doi: 10.3390/jcm10061173. PMID 33799685
- [Derived] Carnevale-Schianca F, Caravelli D, Gallo S, Coha V, D'Ambrosio L, Vassallo E, Fizzotti M, Nesi F, Gioeni L, Berger M, Polo A, Gammaitoni L, Becco P, Giraudo L, Mangioni M, Sangiolo D, Grignani G, Rota-Scalabrini D, Sottile A, Fagioli F, Aglietta M. Post-Transplant Cyclophosphamide and Tacrolimus-Mycophenolate Mofetil Combination Prevents Graft-versus-Host Disease in Allogeneic Peripheral Blood Hematopoietic Cell Transplantation from HLA-Matched Donors. Biol Blood Marrow Transplant. 2017 Mar;23(3):459-466. doi: 10.1016/j.bbmt.2016.12.636. Epub 2016 Dec 27. PMID 28039079